CLINICAL TRIAL: NCT05958017
Title: reSET for the Treatment of Stimulant Use in HIV Clinics: Care Optimization Supporting Treatment Adherence (COSTA)
Acronym: COSTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jose Szapocznik, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20221237; R01DA055563 (NIH)
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Stimulant Use Disorder; People Living With HIV; reSET
Keywords: Substance use; Adherence to Anti-Retroviral Therapy
MeSH Terms: conditions — Substance-Related Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reSET Group (Experimental): Participants in this group will use the reSET mobile app for 12 weeks.
  Interventions: Behavioral: reSET
- Standard of Care Group (Other): Participants in this group will receive standard of care treatment for 12 weeks.
  Interventions: Other: Standard of care

INTERVENTIONS:
Behavioral: reSET — Participants in this group will use a mobile application that delivers treatment for substance use disorder. 31 required and 30 optional modules. Among many topics covered in the modules, some are substance use management, communication, emotion management, relationship skills, HIV/Sexually Transmitted Infections and triggers for risky sex. In the reSET app you will get the chance to earn rewards for two activities: (1) completing a module and (2) providing a negative urine drug screen in exchange for a motivational or monetary prize. You will have 12 weeks to complete as many modules as you like, about 4 modules per week. Each module takes approximately 10-15 min. Every 3-4 days you will meet with the same study team member to provide a urine drug screen from a place comfortable for you (e.g. home) which will be observed and read via Zoom.
  Arms: reSET Group
Other: Standard of care — Participants in this group will receive assistance connecting to an in person community-based outpatient treatment program.
  Arms: Standard of Care Group

SUMMARY:
The purpose of this study is to find out if reSET, an FDA authorized mobile therapeutic, is effective in treating stimulant use disorder and helping keep HIV viral load suppression stable among men who have sex with men who are living with HIV and have a stimulant use disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Identifies as male
2. Reports past year anal intercourse with a male
3. Age 18 or older (reSET is only approved for use with adults)
4. Person living with HIV who is an AIDS Healthcare Foundation (AHF) patient at one of the four metro areas: Atlanta, Dallas/Fort Worth, Fort Lauderdale, Los Angeles
5. Screens positive for a moderate or severe stimulant use disorder in the last 3-months using the MINI
6. Reports that he is not currently in drug treatment
7. Currently has an active antiretroviral therapy prescription and reports < 90% HIV Tx adherence on the 3-item Wilson measure in the past 30 days
8. Can obtain access to stable internet with privacy acceptable to the participant at least twice a week
9. Indicates being able to understand English (reSET is only available in English; can be read or heard)
10. Consents to participation in the study
11. Provides sufficient locator information

Exclusion Criteria:

1. Otherwise eligible participants will be excluded if they appear to display diminished capacity to consent either because of: (a) an apparent inability to provide consent (e.g., cognitive impairment) or (b) apparent severe psychiatric symptoms (e.g., mania, psychosis) that may impair capacity to consent.
2. Persons that meet criteria for prisoner status will be excluded at baseline.
3. Patients who screen positive for moderate to severe opioid use disorder will be excluded from the study because effective pharmacological agents exist for the treatment of this disorder. These patients will be referred to community-based programs that provide specialized treatment for this disorder.
4. Participants will be excluded prior to randomization, if they do not complete at baseline the Time-Line Follow-Back or the laboratory visit.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in days of stimulant use as measured by Timeline FollowBack | 3, 9 and 15 months.
  Number of days of stimulant use as measured by the Timeline FollowBack using the formula: Daily opioid use- the proportion of days of use

SECONDARY OUTCOMES:
Proportion of subjects with viral suppression | 3, 9 and 15 months.
  Changes in RNA viral load. Viral suppression (cv<200copies/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Szapocznik, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No